CLINICAL TRIAL: NCT07113457
Title: Assessing Upper Extremity Function in Chronic Stroke Survivors: Enhancing Neural Recovery With Acute Intermittent Hypoxia
Brief Title: Assessing Upper Extremity Function in Chronic Stroke Survivors Through Acute Intermittent Hypoxia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Zev Rymer, Principal Investigator, Shirley Ryan AbilityLab
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STU00223882; R21NS130367-01 (NIH)
Record Dates: First submitted 2025-07-22; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-07

CONDITIONS: Stroke
Keywords: stroke; hypoxia; spasticity; aih; ultrasound
MeSH Terms: conditions — Stroke; Hypoxia; Muscle Spasticity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hypoxia (Experimental): Participants in this arm will receive approximately 15 bouts of acute intermittent hypoxia. This intervention involves breathing lowered levels of oxygen (similar to being on a tall mountain) for 60 seconds at a time, followed by 60 seconds of room air. Participants will be assessed following the intervention.
  Interventions: Other: Acute Intermittent Hypoxia (AIH)

INTERVENTIONS:
Other: Acute Intermittent Hypoxia (AIH) — This intervention involves breathing lowered levels of oxygen (similar to those experienced on a tall mountain) for 60 seconds at a time. This is immediately followed by 60 seconds of breathing normal room air. These bouts are repeated approximately 15 times. For the intervention, the participant is fitted with a non-rebreathing mask which supplies the two different air levels

SUMMARY:
Here we aim to observe effects of acute intermittent hypoxia in persons who have experienced a single stroke. We have previously shown this technique to be safe and effective at increasing strength in persons with disabilities, and here are aiming to determine the mechanism of how the breathing method modulates motor function.

DETAILED DESCRIPTION:
Here we aim to observe effects of acute intermittent hypoxia in persons who have experienced a single stroke. We have previously shown this technique to be safe and effective at increasing strength in persons with disabilities, and here are aiming to determine the mechanism of how the breathing method modulates motor function.

ELIGIBILITY:
Inclusion Criteria:

* A first time, unilateral, ischemic, hemispheric stroke, confirmed by MRI
* Chedoke stage of hand assessment >= 3
* Ability to open and close affected hand
* Able to understand and communicate in english
* Able to independently consent
* over 6 months post stroke
* Must have a hemoglobin level above 10g/dl
* Must have ability to leave research visit with a compainon/group trasportation
* WOCBP must be comfortable confirming negative pregnancy prior to hypoxia
* Must not be involved in any other research intervention study testing upper extremities

Exclusion Criteria:

* History of prior neurological disorders
* Brain stem or cerebellar stroke; mean Fazekas score rated on initial fluid-attenuated inversion recovery MRI greater than equal to 3
* Severe Aphasisa
* Pre-existing hypoxic pulmonary disease
* Includes positive Covid-pneumonia diagnosis within 1 year of screening visit
* Severe hypertension (>160/100)
* Any ischemic cardiac disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Joint Force Measurement | 30 minutes following intervention
  The KAIST Upper Limb Synergy Investigation System (KULSIS) will be utilized. KULSIS was developed in collaboration with Neuro-
  Figure 1: Design of the KULSIS Rehabilitation Engineering Lab at Korea Advanced Institute of Science and Technology, South Korea (Figure 1). It comprises a modular hand and wrist attachment, which connects to a linear actuator. To construct the linear actuator, ball-screw type linear motion module (RS-075N-Z05PR, Robostar, South Korea) was combined with a 100 W AC servo motor (SGM7J-01AFD2C, Yaskawa, Japan). The linear actuator has stroke range of 400 mm, which is ample for adjusting the position of modular hand or wrist attachment to the participant's upper arm before the outcome assessment. Once adjusted, the power of linear actuator will be turned off to fix the position.
  A six degrees of freedom (DOF) Force/Torque sensor (Series Delta, ATI-Inc. Apex, NC, USA) is positioned between the module and the linear actuator to measure the force and torque applie

SECONDARY OUTCOMES:
Stretch reflex measurement: | 30 minutes following intervention
  Stretch reflex thresholds will be assessed using a custom-designed tendon tapper system (Figure 2.A) based on a Linmot® linear motor (Linmot S.A., Spreitenbach, Switzerland). This system includes a stator and slider with integrated position sensing via a Hall effect sensor, ensuring precise control of tendon indentations and taps. The motor is mounted on a micrometer-driven positioner (Velmex, Bloomfield, NY, USA) for reliable placement of the tapper on the biceps brachii tendon. A multiaxial load cell (Series Nano17, ATI Industrial Automation, Apex, NC, USA) is attached at the tapping end to record applied forces and the resultant reflex responses. Additionally, the tendon tapper integrates a wireless ultrasound device(Figure 2.B) at its tip to provide real-time transverse imaging of the tissue composition surrounding the distal biceps tendon. The ultrasound device features an image resolution of 384 pixels (width) by 400-600 pixels (depth), corresponding to a physical size of 38.4 m
Surface EMG measurement | 30 minutes following intervention
  Surface EMG signals will be recorded using two systems to capture muscle activity during isometric contractions. The Bagnoli-8 EMG system (Delsys Inc, Boston, MA, USA), equipped with standard wired bipolar surface EMG electrodes, will provide localized muscle activity measurements. Additionally, high-density surface EMG (HDsEMG) recordings will be conducted using a 128-channel Refa system (TMSi; Oldenzaal, NL) with an 8×8 electrode grid (8.5 mm inter-electrode distance) to map spatially distributed muscle activity with high resolution (Figure 3). These complementary systems will allow a comprehensive assessment of muscle activation patterns during the study.
EKG | Continuously throughout intervention up to 30 minutes post intervention
  Standard bedside monitoring- a 2-lead tracing to identify dysrhythmias. EKG to be performed throughout hypoxia administration. 12 lead ECG to be performed at visit 1 at resting state with no other ongoing activities
Symptom Checklist | at each time point: 2, 6, 14, 24 and 30mins from the beginning of the hypoxia session.
  A simple yes/no subjective checklist will be asked and repeated to the subject. Specifically: Chest pain, Shortness of breath, Light headedness, neck pain, dizziness, arm pain, sweaty, sensory changes, increased weakness

CONTACTS AND LOCATIONS:
Overall Officials: William Z Rymer, MD, PhD, Principal Investigator — Shirley Ryan AbilityLab

IPD SHARING:
Plan to Share IPD: Yes
De-identified results will be shared upon request
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Within 1 year of study conclusions
Access Criteria: Study staff only has access to the full data sets and will provide relevant data upon request